CLINICAL TRIAL: NCT03597438
Title: Mitochondrial Targeted Biofuels as Countermeasures Against Chemical Threats
Brief Title: National CounterACT Initiative
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-015056; 1R21NS103826-01 (NIH)
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Mitochondrial Alteration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: patients scheduled for elective surgery who are patients either as an inpatient or arriving to the hospital on the day of scheduled surgery
- Volunteer: Volunteers who are employees, trainees and students at the Children's Hospital of Philadelphia (CHOP) will be introduced to the study via an informational study flyer to determine eligibility and desire to participate in the study

SUMMARY:
The purpose of the study is to determine in vitro effects on mitochondrial function of selected chemical agents in human cells, and assess the capability of a cell-permeable succinate prodrug to attenuate toxic effects The project aims at repurposing this recent pharmaceutical discovery, currently being developed for treatment of toxic exposure, for an expanded indication to treat chemically induced mitochondrial toxicity.

DETAILED DESCRIPTION:
The study duration per subject will be approximately 15 minutes to complete the one time blood collection.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Males or females age greater or equal 2 years of age
2. Weight greater or equal to 10 kg
3. Parental/guardian permission (informed consent) and if appropriate, child assent.

Patient Exclusion Criteria:

1. Known primary mitochondrial disorder.
2. Use of an investigational drug within 30 days prior to enrollment.
3. Parents/guardians or subjects who in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Volunteer Inclusion Criteria

1. Males or females > 18 years of age
2. Employee, trainee, or student informed consent

Volunteer Exclusion Criteria:

1. Prior enrollment in this study.
2. Known primary mitochondrial disorder.
3. Use of an investigational drug within 30 days prior to enrollment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for elective surgery will be screened for eligibility. Volunteers who are employees, trainees, and students will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Attenuation by the succinate prodrug of toxin-induced decrease in mitochondrial respiration. | by end of 2018
  Data will be assessed using 2-tailed Student's t-test. Dose-response curves for respiration will be made for each toxin and IC50 calculated. In case of difficulties in demonstrating acute toxicity of chemical agents, dose-titration experiments and long-term incubation (up to 24 hours) will be performed

SECONDARY OUTCOMES:
Attenuation of toxin-induced decrease in mitochondrial membrane potential and attenuate lactate production by the succinate prodrug. | by end of 2018
  Data will be assessed using 2-tailed Student's t-test. Dose-response curves for respiration will be made for each toxin and IC50 calculated. In case of difficulties in demonstrating acute toxicity of chemical agents, dose-titration experiments and long-term incubation (up to 24 h) will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Todd J Kilbaugh, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeevaratnam K, Vidya S, Vaidyanathan CS. In vitro and in vivo effect of methyl isocyanate on rat liver mitochondrial respiration. Toxicol Appl Pharmacol. 1992 Dec;117(2):172-9. doi: 10.1016/0041-008x(92)90234-j. PMID 1471148
- [Background] Ehinger JK, Piel S, Ford R, Karlsson M, Sjovall F, Frostner EA, Morota S, Taylor RW, Turnbull DM, Cornell C, Moss SJ, Metzsch C, Hansson MJ, Fliri H, Elmer E. Cell-permeable succinate prodrugs bypass mitochondrial complex I deficiency. Nat Commun. 2016 Aug 9;7:12317. doi: 10.1038/ncomms12317. PMID 27502960
- [Background] Degli Esposti M. Inhibitors of NADH-ubiquinone reductase: an overview. Biochim Biophys Acta. 1998 May 6;1364(2):222-35. doi: 10.1016/s0005-2728(98)00029-2. PMID 9593904
- [Background] Mesnage R, Arno M, Costanzo M, Malatesta M, Seralini GE, Antoniou MN. Transcriptome profile analysis reflects rat liver and kidney damage following chronic ultra-low dose Roundup exposure. Environ Health. 2015 Aug 25;14:70. doi: 10.1186/s12940-015-0056-1. PMID 26302742
- [Background] Friedrich T, van Heek P, Leif H, Ohnishi T, Forche E, Kunze B, Jansen R, Trowitzsch-Kienast W, Hofle G, Reichenbach H, et al. Two binding sites of inhibitors in NADH: ubiquinone oxidoreductase (complex I). Relationship of one site with the ubiquinone-binding site of bacterial glucose:ubiquinone oxidoreductase. Eur J Biochem. 1994 Jan 15;219(1-2):691-8. doi: 10.1111/j.1432-1033.1994.tb19985.x. PMID 8307034
- [Background] Lim S, Ahn SY, Song IC, Chung MH, Jang HC, Park KS, Lee KU, Pak YK, Lee HK. Chronic exposure to the herbicide, atrazine, causes mitochondrial dysfunction and insulin resistance. PLoS One. 2009;4(4):e5186. doi: 10.1371/journal.pone.0005186. Epub 2009 Apr 13. PMID 19365547
- [Background] Hase Y, Tatsuno M, Nishi T, Kataoka K, Kabe Y, Yamaguchi Y, Ozawa N, Natori M, Handa H, Watanabe H. Atrazine binds to F1F0-ATP synthase and inhibits mitochondrial function in sperm. Biochem Biophys Res Commun. 2008 Feb 1;366(1):66-72. doi: 10.1016/j.bbrc.2007.11.107. Epub 2007 Dec 4. PMID 18060860
- [Background] Hollingworth RM, Ahammadsahib KI, Gadelhak G, McLaughlin JL. New inhibitors of complex I of the mitochondrial electron transport chain with activity as pesticides. Biochem Soc Trans. 1994 Feb;22(1):230-3. doi: 10.1042/bst0220230. No abstract available. PMID 8206238
- [Background] Satoh T, Miyoshi H, Sakamoto K, Iwamura H. Comparison of the inhibitory action of synthetic capsaicin analogues with various NADH-ubiquinone oxidoreductases. Biochim Biophys Acta. 1996 Jan 11;1273(1):21-30. doi: 10.1016/0005-2728(95)00131-x. PMID 8573592
- [Background] Gassner B, Wuthrich A, Scholtysik G, Solioz M. The pyrethroids permethrin and cyhalothrin are potent inhibitors of the mitochondrial complex I. J Pharmacol Exp Ther. 1997 May;281(2):855-60. PMID 9152394
- [Background] Gunnell D, Eddleston M, Phillips MR, Konradsen F. The global distribution of fatal pesticide self-poisoning: systematic review. BMC Public Health. 2007 Dec 21;7:357. doi: 10.1186/1471-2458-7-357. PMID 18154668
- [Background] Bus JS, Gibson JE. Paraquat: model for oxidant-initiated toxicity. Environ Health Perspect. 1984 Apr;55:37-46. doi: 10.1289/ehp.845537. PMID 6329674
- [Background] Tawara T, Fukushima T, Hojo N, Isobe A, Shiwaku K, Setogawa T, Yamane Y. Effects of paraquat on mitochondrial electron transport system and catecholamine contents in rat brain. Arch Toxicol. 1996;70(9):585-9. doi: 10.1007/s002040050316. PMID 8831909
- [Background] Eckerman I. THE BHOPAL SAGA: Universities Press (India); 2005.